CLINICAL TRIAL: NCT04839159
Title: Prospective Clinical Study on Early Inflammatory, Cell Adhesion and Hemostatic Plasmatic Markers of Endothelial Dysfunction in Children With Sickle Cell Disease (SCD)
Brief Title: Study of Biological Markers in Children With Sickle Cell Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Queen Fabiola Children's University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P2012/SCD1
Record Dates: First submitted 2018-07-11; First posted 2021-04-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Sickle Cell Disease
Keywords: Sickle cell disease, children, thrombin generation, inflammation, cytokines, adhesion molecules, plasmatic markers, coagulation
MeSH Terms: conditions — Anemia, Sickle Cell; Inflammation; Thrombosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SCD Patient (Experimental)
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Blood sampling at the age of 6 and 12 months, 2-3-4 years
Other: Blood sampling — Blood sampling before any new sickle cell disease treatment as determined by a physician according to the standard of care to which the hospital adheres

SUMMARY:
Sickle cell disease is associated with significant morbi-mortality hence the interest in an early and targeted care. At present, there is no plasmatic marker able to identify infants at higher risk of developping severe complications later in life. However, recent studies have demonstrated a correlation between certain complications of the disease and biomarkers of the endothelial dysfunction characterizing it.

Investigators prospectively followed a cohort of children diagnosed with SCD through the universal neonatal screening using inflammatory and haemostatic plasmatic markers to study their annual evolution. Investigators then will evaluate potential associations between these biological markers and the occurrence of SCD related complications. A secondary objective of this study is to evaluate the repercussions of therapeutic intervention on these markers.

.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged less than 6 months
* Sickle cell syndrome SS, Sβthal or SC confirmed by hemoglobin electrophoresis
* Subjects legal representatives must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to let participate their child in the study

Exclusion Criteria:

* Congenital abnormality other than sickle cell disease except for a glucose-6-phosphate-deshydrogenase
* Prematurity
* Initiation of the following therapies before enrollment: chronic transfusion regimen or bone marrow transplantation

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2012-05-10 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Plasmatic levels of IL-6 at 12 months of age | 12 months of age
  Measurement of plasmatic levels of IL-6 (fg/mL) by flow cytometric assay

SECONDARY OUTCOMES:
Plasmatic levels of IL-6 at 6 months of age | 6 months of age
  Measurement of plasmatic levels of IL-6 (fg/mL) by flow cytometric assay
Plasmatic levels of IL-6 at 2 years of age | 2 years of age
  Measurement of plasmatic levels of IL-6 (fg/mL) by flow cytometric assay
Plasmatic levels of IL-6 at 3 years of age | 3 years of age
  Measurement of plasmatic levels of IL-6 (fg/mL) by flow cytometric assay
Plasmatic levels of IL-6 at 4 years of age | 4 years of age
  Measurement of plasmatic levels of IL-6 (fg/mL) by flow cytometric assay
Plasmatic levels of IL-6 before the introduction of any new sickle cell disease treatment as determined by a physician according to the standard of care to which the hospital adheres | Before the introduction of any new sickle cell disease treatment
  Measurement of plasmatic levels of IL-6 (fg/mL) by flow cytometric assay
Plasmatic levels of IL-1ß at 6 months of age | 6 months of age
  Measurement of plasmatic levels of IL-1ß (fg/mL) by flow cytometric assay
Plasmatic levels of IL-1ß at 12 months of age | 12 months of age
  Measurement of plasmatic levels of IL-1ß (fg/mL) by flow cytometric assay
Plasmatic levels of IL-1ß at 2 years of age | 2 years of age
  Measurement of plasmatic levels of IL-1ß (fg/mL) by flow cytometric assay
Plasmatic levels of IL-1ß at 3 years of age | 3 years of age
  Measurement of plasmatic levels of IL-1ß (fg/mL) by flow cytometric assay
Plasmatic levels of IL-1ß at 4 years of age | 4 years of age
  Measurement of plasmatic levels of IL-1ß (fg/mL) by flow cytometric assay
Plasmatic levels of IL-1ß before the introduction of any new sickle cell disease treatment as determined by a physician according to the standard of care to which the hospital adheres | Before the introduction of any new sickle cell disease treatment
  Measurement of plasmatic levels of IL-1ß (fg/mL) by flow cytometric assay
Plasmatic levels of IL-8 at 6 months of age | 6 months of age
  Measurement of plasmatic levels of IL-8 (fg/mL) by flow cytometric assay
Plasmatic levels of IL-8 at 12 months of age | 12 months of age
  Measurement of plasmatic levels of IL-8 (fg/mL) by flow cytometric assay
Plasmatic levels of IL-8 at 2 years of age | 2 years of age
  Measurement of plasmatic levels of IL-8 (fg/mL) by flow cytometric assay
Plasmatic levels of IL-8 at 3 years of age | 3 years of age
  Measurement of plasmatic levels of IL-8 (fg/mL) by flow cytometric assay
Plasmatic levels of IL-8 at 4 years of age | 4 years of age
  Measurement of plasmatic levels of IL-8 (fg/mL) by flow cytometric assay
Plasmatic levels of IL-8 before the introduction of any new sickle cell disease treatment as determined by a physician according to the standard of care to which the hospital adheres | Before the introduction of any new sickle cell disease treatment
  Measurement of plasmatic levels of IL-8 (fg/mL) by flow cytometric assay
Plasmatic levels of IL-10 at 6 months of age | 6 months of age
  Measurement of plasmatic levels of IL-10 (fg/mL) by flow cytometric assay
Plasmatic levels of IL-10 at 12 months of age | 12 months of age
  Measurement of plasmatic levels of IL-10 (fg/mL) by flow cytometric assay
Plasmatic levels of IL-10 at 2 years of age | 2 years of age
  Measurement of plasmatic levels of IL-10 (fg/mL) by flow cytometric assay
Plasmatic levels of IL-10 at 3 years of age | 3 years of age
  Measurement of plasmatic levels of IL-10 (fg/mL) by flow cytometric assay
Plasmatic levels of IL-10 at 4 years of age | 4 years of age
  Measurement of plasmatic levels of IL-10 (fg/mL) by flow cytometric assay
Plasmatic levels of IL-10 before the introduction of any new sickle cell disease treatment as determined by a physician according to the standard of care to which the hospital adheres | Before the introduction of any new sickle cell disease treatment
  Measurement of plasmatic levels of IL-10 (fg/mL) by flow cytometric assay
Plasmatic levels of IL-12 at 6 months of age | 6 months of age
  Measurement of plasmatic levels of IL-12 (fg/mL) by flow cytometric assay
Plasmatic levels of IL-12 at 12 months of age | 12 months of age
  Measurement of plasmatic levels of IL-12 (fg/mL) by flow cytometric assay
Plasmatic levels of IL-12 at 2 years of age | 2 years of age
  Measurement of plasmatic levels of IL-12 (fg/mL) by flow cytometric assay
Plasmatic levels of IL-12 at 3 years of age | 3 years of age
  Measurement of plasmatic levels of IL-12 (fg/mL) by flow cytometric assay
Plasmatic levels of IL-12 at 4 years of age | 4 years of age
  Measurement of plasmatic levels of IL-12 (fg/mL) by flow cytometric assay
Plasmatic levels of IL-12 before the introduction of any new sickle cell disease treatment as determined by a physician according to the standard of care to which the hospital adheres | Before the introduction of any new sickle cell disease treatment
  Measurement of plasmatic levels of IL-12 (fg/mL) by flow cytometric assay
Plasmatic levels of TNF alpha at 6 months of age | 6 months of age
  Measurement of plasmatic levels of TNF alpha (fg/mL) by flow cytometric assay
Plasmatic levels of TNF alpha at 12 months of age | 12 months of age
  Measurement of plasmatic levels of TNF alpha (fg/mL) by flow cytometric assay
Plasmatic levels of TNF alpha at 2 years of age | 2 years of age
  Measurement of plasmatic levels of TNF alpha (fg/mL) by flow cytometric assay
Plasmatic levels of TNF alpha at 3 years of age | 3 years of age
  Measurement of plasmatic levels of TNF alpha (fg/mL) by flow cytometric assay
Plasmatic levels of TNF alpha at 4 years of age | 4 years of age
  Measurement of plasmatic levels of TNF alpha (fg/mL) by flow cytometric assay
Plasmatic levels of TNF alpha before the introduction of any new sickle cell disease treatment as determined by a physician according to the standard of care to which the hospital adheres | Before the introduction of any new sickle cell disease treatment
  Measurement of plasmatic levels of TNF alpha (fg/mL) by flow cytometric assay
Plasmatic levels of ICAM-1 at 6 months of age | 6 months of age
  Measurement of plasmatic levels of ICAM-1 (pg/mL) by flow cytometric assay
Plasmatic levels of ICAM-1 at 12 months of age | 12 months of age
  Measurement of plasmatic levels of ICAM-1 (pg/mL) by flow cytometric assay
Plasmatic levels of ICAM-1 at 2 years of age | 2 years of age
  Measurement of plasmatic levels of ICAM-1 (pg/mL) by flow cytometric assay
Plasmatic levels of ICAM-1 at 3 years of age | 3 years of age
  Measurement of plasmatic levels of ICAM-1 (pg/mL) by flow cytometric assay
Plasmatic levels of ICAM-1 at 4 years of age | 4 years of age
  Measurement of plasmatic levels of ICAM-1 (pg/mL) by flow cytometric assay
Plasmatic levels of ICAM-1 before the introduction of any new sickle cell disease treatment as determined by a physician according to the standard of care to which the hospital adheres | Before the introduction of any new sickle cell disease treatment
  Measurement of plasmatic levels of ICAM-1 (pg/mL) by flow cytometric assay
Plasmatic levels of VCAM-1 at 6 months of age | 6 months of age
  Measurement of plasmatic levels of VCAM-1 (pg/mL) by flow cytometric assay
Plasmatic levels of VCAM-1 at 12 months of age | 12 months of age
  Measurement of plasmatic levels of VCAM-1 (pg/mL) by flow cytometric assay
Plasmatic levels of VCAM-1 at 2 years of age | 2 years of age
  Measurement of plasmatic levels of VCAM-1 (pg/mL) by flow cytometric assay
Plasmatic levels of VCAM-1 at 3 years of age | 3 years of age
  Measurement of plasmatic levels of VCAM-1 (pg/mL) by flow cytometric assay
Plasmatic levels of VCAM-1 at 4 years of age | 4 years of age
  Measurement of plasmatic levels of VCAM-1 (pg/mL) by flow cytometric assay
Plasmatic levels of VCAM-1 before the introduction of any new sickle cell disease treatment as determined by a physician according to the standard of care to which the hospital adheres | Before the introduction of any new sickle cell disease treatment
  Measurement of plasmatic levels of VCAM-1 (pg/mL) by flow cytometric assay
Plasmatic VCAM-1 levels after in vitro stimulation with LPS | Plasmatic level of VCAM-1 after in vitro stimulation with LPS
  Measurement of plasmatic levels of VCAM-1 (pg/mL) by flow cytometric assay after in vitro stimulation with LPS
Plasmatic levels of E-selectine at 6 months of age | 6 months of age
  Measurement of plasmatic levels of E-selectine (pg/mL) by flow cytometric assay
Plasmatic levels of E-selectine at 12 months of age | 12 months of age
  Measurement of plasmatic levels of E-selectine (pg/mL) by flow cytometric assay
Plasmatic levels of E-selectine at 2 years of age | 2 years of age
  Measurement of plasmatic levels of E-selectine (pg/mL) by flow cytometric assay
Plasmatic levels of E-selectine at 3 years of age | 3 years of age
  Measurement of plasmatic levels of E-selectine (pg/mL) by flow cytometric assay
Plasmatic levels of E-selectine at 4 years of age | 4 years of age
  Measurement of plasmatic levels of E-selectine (pg/mL) by flow cytometric assay
Plasmatic levels of E-selectine before the introduction of any new sickle cell disease treatment as determined by a physician according to the standard of care to which the hospital adheres | Before the introduction of any new sickle cell disease treatment
  Measurement of plasmatic levels of E-selectine (pg/mL) by flow cytometric assay
Plasmatic levels of P-selectine at 6 months of age | 6 months of age
  Measurement of plasmatic levels of P-selectine (pg/mL) by flow cytometric assay
Plasmatic levels of P-selectine at 12 months of age | 12 months of age
  Measurement of plasmatic levels of P-selectine (pg/mL) by flow cytometric assay
Plasmatic levels of P-selectine at 2 years of age | 2 years of age
  Measurement of plasmatic levels of P-selectine (pg/mL) by flow cytometric assay
Plasmatic levels of P-selectine at 3 years of age | 3 years of age
  Measurement of plasmatic levels of P-selectine (pg/mL) by flow cytometric assay
Plasmatic levels of P-selectine at 4 years of age | 4 years of age
  Measurement of plasmatic levels of P-selectine (pg/mL) by flow cytometric assay
Plasmatic levels of P-selectine before the introduction of any new sickle cell disease treatment as determined by a physician according to the standard of care to which the hospital adheres | Before the introduction of any new sickle cell disease treatment
  Measurement of plasmatic levels of P-selectine (pg/mL) by flow cytometric assay
Plasmatic levels of Vascular Endothelial Growth Factor (VEGF) at 6 months of age | 6 months of age
  Measurement of plasmatic levels of VEGF (pg/mL) by flow cytometric assay
Plasmatic levels of Vascular Endothelial Growth Factor (VEGF) at 12 months of age | 12 months of age
  Measurement of plasmatic levels of VEGF (pg/mL) by flow cytometric assay
Plasmatic levels of Vascular Endothelial Growth Factor (VEGF) at 2 years of age | 2 years of age
  Measurement of plasmatic levels of VEGF (pg/mL) by flow cytometric assay
Plasmatic levels of Vascular Endothelial Growth Factor (VEGF) at 3 years of age | 3 years of age
  Measurement of plasmatic levels of VEGF (pg/mL) by flow cytometric assay
Plasmatic levels of Vascular Endothelial Growth Factor (VEGF) at 4 years of age | 4 years of age
  Measurement of plasmatic levels of VEGF (pg/mL) by flow cytometric assay
Plasmatic levels of VEGF before the introduction of any new sickle cell disease treatment as determined by a physician according to the standard of care to which the hospital adheres | Before the introduction of any new sickle cell disease treatment
  Measurement of plasmatic levels of VEGF (pg/mL) by flow cytometric assay
Lag time parameter in thrombin generation assay at 6 months of age | 6 months of age
  Measurement of lag time (minutes) parameter of thrombin generation in platelet poor plasma using the Calibrated Automated Thrombogram (CAT®) method.
Lag time parameter in thrombin generation assay at 12 months of age | 12 months of age
  Measurement of lag time (minutes) parameter of thrombin generation in platelet poor plasma using the Calibrated Automated Thrombogram (CAT®) method.
Lag time parameter in thrombin generation assay at 2 years of age | 2 years of age
  Measurement of lag time (minutes) parameter of thrombin generation in platelet poor plasma using the Calibrated Automated Thrombogram (CAT®) method.
Lag time parameter in thrombin generation assay at 3 years of age | 3 years of age
  Measurement of lag time (minutes) parameter of thrombin generation in platelet poor plasma using the Calibrated Automated Thrombogram (CAT®) method.
Lag time parameter in thrombin generation assay at 4 years of age | 4 years of age
  Measurement of lag time (minutes) parameter of thrombin generation in platelet poor plasma using the Calibrated Automated Thrombogram (CAT®) method.
Lag time parameter in thrombin generation assay before the introduction of any new sickle cell disease treatment as determined by a physician according to the standard of care to which the hospital adheres | Before the introduction of any new sickle cell disease treatment
  Measurement of lag time (minutes) parameter of thrombin generation in platelet poor plasma using the Calibrated Automated Thrombogram (CAT®) method.
Peak height parameter in thrombin generation assay at 6 months of age | 6 months of age
  Measurement of peak height (nM) parameter of thrombin generation in platelet poor plasma using the Calibrated Automated Thrombogram (CAT®) method.
Peak height parameter in thrombin generation assay at 12 months of age | 12 months of age
  Measurement of peak height (nM) parameter of thrombin generation in platelet poor plasma using the Calibrated Automated Thrombogram (CAT®) method.
Peak height parameter in thrombin generation assay at 2 years of age | 2 years of age
  Measurement of peak height (nM) parameter of thrombin generation in platelet poor plasma using the Calibrated Automated Thrombogram (CAT®) method.
Peak height parameter in thrombin generation assay at 3 years of age | 3 years of age
  Measurement of peak height (nM) parameter of thrombin generation in platelet poor plasma using the Calibrated Automated Thrombogram (CAT®) method.
Peak height parameter in thrombin generation assay at 4 years of age | 4 years of age
  Measurement of peak height (nM) parameter of thrombin generation in platelet poor plasma using the Calibrated Automated Thrombogram (CAT®) method.
Peak height parameter in thrombin generation assay before the introduction of any new sickle cell disease treatment as determined by a physician according to the standard of care to which the hospital adheres | Before the introduction of any new sickle cell disease treatment
  Measurement of peak height (nM) parameter of thrombin generation in platelet poor plasma using the Calibrated Automated Thrombogram (CAT®) method.
Time to peak parameter in thrombin generation assay at 6 months of age | 6 months of age
  Measurement of time to peak (minutes) parameter of thrombin generation in platelet poor plasma using the Calibrated Automated Thrombogram (CAT®) method
Time to peak parameter in thrombin generation assay at 12 months of age | 12 months of age
  Measurement of time to peak (minutes) parameter of thrombin generation in platelet poor plasma using the Calibrated Automated Thrombogram (CAT®) method
Time to peak parameter in thrombin generation assay at 2 years of age | 2 years of age
  Measurement of time to peak (minutes) parameter of thrombin generation in platelet poor plasma using the Calibrated Automated Thrombogram (CAT®) method
Time to peak parameter in thrombin generation assay at 3 years of age | 3 years of age
  Measurement of time to peak (minutes) parameter of thrombin generation in platelet poor plasma using the Calibrated Automated Thrombogram (CAT®) method
Time to peak parameter in thrombin generation assay at 4 years of age | 4 years of age
  Measurement of time to peak (minutes) parameter of thrombin generation in platelet poor plasma using the Calibrated Automated Thrombogram (CAT®) method
Time to peak parameter in thrombin generation assay before the introduction of any new sickle cell disease treatment as determined by a physician according to the standard of care to which the hospital adheres | Before the introduction of any new sickle cell disease treatment
  Measurement of time to peak (minutes) parameter of thrombin generation in platelet poor plasma using the Calibrated Automated Thrombogram (CAT®) method
Endogenous thrombin potential parameter in thrombin generation assay at 6 months of age | 6 months of age
  Measurement of endogenous thrombin potential (nM x minutes) parameter of thrombin generation in platelet poor plasma using the Calibrated Automated Thrombogram (CAT®) method.
Endogenous thrombin potential parameter in thrombin generation assay at 12 months of age | 12 months of age
  Measurement of endogenous thrombin potential (nM x minutes) parameter of thrombin generation in platelet poor plasma using the Calibrated Automated Thrombogram (CAT®) method.
Endogenous thrombin potential parameter in thrombin generation assay at 2 years of age | 2 years of age
  Measurement of endogenous thrombin potential (nM x minutes) parameter of thrombin generation in platelet poor plasma using the Calibrated Automated Thrombogram (CAT®) method.
Endogenous thrombin potential parameter in thrombin generation assay at 3 years of age | 3 years of age
  Measurement of endogenous thrombin potential (nM x minutes) parameter of thrombin generation in platelet poor plasma using the Calibrated Automated Thrombogram (CAT®) method.
Endogenous thrombin potential parameter in thrombin generation assay at 4 years of age | 4 years of age
  Measurement of endogenous thrombin potential (nM x minutes) parameter of thrombin generation in platelet poor plasma using the Calibrated Automated Thrombogram (CAT®) method.
Endogenous thrombin potential parameter in thrombin generation assay before the introduction of any new sickle cell disease treatment as determined by a physician according to the standard of care to which the hospital adheres | before the introduction of any new sickle cell disease treatment
  Measurement of endogenous thrombin potential (nM x minutes) parameter of thrombin generation in platelet poor plasma using the Calibrated Automated Thrombogram (CAT®) method.
Plasmatic levels of Factor VIII at 6 months of age | 6 months of age
  Measurement of plasmatic levels of Factor VIII by flow cytometric assay
Plasmatic levels of Factor VIII at 12 months of age | 12 months of age
  Measurement of plasmatic levels of Factor VIII by flow cytometric assay
Plasmatic levels of Factor VIII at 2 years of age | 2 years of age
  Measurement of plasmatic levels of Factor VIII by flow cytometric assay
Plasmatic levels of Factor VIII at 3 years of age | 3 years of age
  Measurement of plasmatic levels of Factor VIII by flow cytometric assay
Plasmatic levels of Factor VIII at 4 years of age | 4 years of age
  Measurement of plasmatic levels of Factor VIII by flow cytometric assay
Plasmatic levels of Factor VIII before the introduction of any new sickle cell disease treatment as determined by a physician according to the standard of care to which the hospital adheres | Before the introduction of any new sickle cell disease treatment
  Measurement of plasmatic levels of Factor VIII by flow cytometric assay

CONTACTS AND LOCATIONS:
Overall Officials: Bushra Zucca, MD, Principal Investigator — Queen Fabiola Children's University Hospital
Locations (3):
- Belgium (3):
  - CHU Saint Pierre, Brussels
  - Hôpital Universitaire Des Enfants Reine Fabiola, Brussels
  - HIS - Site Etterbeek-Ixelles, Brussels

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ware RE, de Montalembert M, Tshilolo L, Abboud MR. Sickle cell disease. Lancet. 2017 Jul 15;390(10091):311-323. doi: 10.1016/S0140-6736(17)30193-9. Epub 2017 Feb 1. PMID 28159390
- [Background] Gulbis B, Cotton F, Ferster A, Ketelslegers O, Dresse MF, Ronge-Collard E, Minon JM, Le PQ, Vertongen F. Neonatal haemoglobinopathy screening in Belgium. J Clin Pathol. 2009 Jan;62(1):49-52. doi: 10.1136/jcp.2008.060517. PMID 19103861
- [Background] Ballas SK, Lieff S, Benjamin LJ, Dampier CD, Heeney MM, Hoppe C, Johnson CS, Rogers ZR, Smith-Whitley K, Wang WC, Telen MJ; Investigators, Comprehensive Sickle Cell Centers. Definitions of the phenotypic manifestations of sickle cell disease. Am J Hematol. 2010 Jan;85(1):6-13. doi: 10.1002/ajh.21550. PMID 19902523
- [Background] Horan J, Lerner N. Prediction of adverse outcomes in children with sickle cell disease. N Engl J Med. 2000 May 25;342(21):1612-3. doi: 10.1056/NEJM200005253422114. No abstract available. PMID 10841686
- [Background] Miller ST, Sleeper LA, Pegelow CH, Enos LE, Wang WC, Weiner SJ, Wethers DL, Smith J, Kinney TR. Prediction of adverse outcomes in children with sickle cell disease. N Engl J Med. 2000 Jan 13;342(2):83-9. doi: 10.1056/NEJM200001133420203. PMID 10631276
- [Background] Quinn CT, Lee NJ, Shull EP, Ahmad N, Rogers ZR, Buchanan GR. Prediction of adverse outcomes in children with sickle cell anemia: a study of the Dallas Newborn Cohort. Blood. 2008 Jan 15;111(2):544-8. doi: 10.1182/blood-2007-07-100719. Epub 2007 Oct 1. PMID 17909076
- [Background] Gladwin MT, Vichinsky E. Pulmonary complications of sickle cell disease. N Engl J Med. 2008 Nov 20;359(21):2254-65. doi: 10.1056/NEJMra0804411. No abstract available. PMID 19020327
- [Background] Charrin E, Ofori-Acquah SF, Nader E, Skinner S, Connes P, Pialoux V, Joly P, Martin C. Inflammatory and oxidative stress phenotypes in transgenic sickle cell mice. Blood Cells Mol Dis. 2016 Nov;62:13-21. doi: 10.1016/j.bcmd.2016.10.020. Epub 2016 Oct 28. PMID 27835777
- [Background] Sarray S, Saleh LR, Lisa Saldanha F, Al-Habboubi HH, Mahdi N, Almawi WY. Serum IL-6, IL-10, and TNFalpha levels in pediatric sickle cell disease patients during vasoocclusive crisis and steady state condition. Cytokine. 2015 Mar;72(1):43-7. doi: 10.1016/j.cyto.2014.11.030. Epub 2015 Jan 5. PMID 25569375
- [Background] Hoppe C, Klitz W, Noble J, Vigil L, Vichinsky E, Styles L. Distinct HLA associations by stroke subtype in children with sickle cell anemia. Blood. 2003 Apr 1;101(7):2865-9. doi: 10.1182/blood-2002-09-2791. Epub 2002 Nov 27. PMID 12517810
- [Background] Garrido VT, Proenca-Ferreira R, Dominical VM, Traina F, Bezerra MA, de Mello MR, Colella MP, Araujo AS, Saad ST, Costa FF, Conran N. Elevated plasma levels and platelet-associated expression of the pro-thrombotic and pro-inflammatory protein, TNFSF14 (LIGHT), in sickle cell disease. Br J Haematol. 2012 Sep;158(6):788-97. doi: 10.1111/j.1365-2141.2012.09218.x. Epub 2012 Jul 6. PMID 22775554